CLINICAL TRIAL: NCT06444919
Title: Capsaicin in Digital Osteoarthritis Versus Control : a Randomized Study
Brief Title: Capsaicin in Digital Osteoarthritis Versus Control
Acronym: CADOR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC IR 2022 MATHIEU; 2024-511159-16-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis Hand; Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Capsaicin; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsaicin 8% (Experimental): patch 179 mg, 30 min
  Interventions: Drug: Capsaicin 179 Mg Cutaneous Patch
- Capsaicin 0.04% (Sham Comparator): patch low dose, 30 min
  Interventions: Drug: Capsaicine low dose 0.04 %

INTERVENTIONS:
Drug: Capsaicin 179 Mg Cutaneous Patch — patch application for 30 minutes on the painful fingers.
  Other Names: QUTENZA
  Arms: Capsaicin 8%
Drug: Capsaicine low dose 0.04 % — patch application for 30 minutes on the painful fingers. the low-dose patch has a similar appearance to the active patch. It allows you to keep the blind, because it also causes reactions at the capsaicin application site (erythema, burning).
  Other Names: control treatment
  Arms: Capsaicin 0.04%

SUMMARY:
The objective of this multicentric, randomized controlled double-blind clinical trial is to demonstrate the efficacy of transdermal application of capsaicin in patients with painful digital osteoarthritis with a neuropathic pain component.

Participants will receive either a transdermal patch of capsaicin 179 mg (8%) or the control treatment (capsaicin 0.04%).

Researchers will compare the intensity of pain in the fingers at day 60 in the capsaicin 8% group versus capsaicin 0.04% (control arm)

DETAILED DESCRIPTION:
Visit 0 : Screening visit (D0 - 30 days): Screen for eligibility

Visit 1 :Inclusion visit (D0): Randomization and blinded patch application of capsaicin 8% or 0.04%

Visit 2: Follow-up visit 1 (D60 + 7 days): Assessment +/- Patch renewal. Patients with finger pain still greater than 4/10 may receive an open application of a capsaicin 8%

Visit 3:Follow-up visit 2 (D120 +/- 7 days): Final assessment.

For the duration of the study, the patient will record in a notebook: analgesics, anti-inflammatories, corticoids and daily hand pain VAS.

Blood samples will be taken at V1 and V2 for subsequent measurement of pro-inflammatory cytokines (IL6, IL8, TNFa) and markers of cartilage degradation, in order to build up a serum library.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of digital osteoarthritis fulfilling the American College of Rheumatology criteria;
* Presence of finger pain of ≥ 40 mm on a visual analogue scale (VAS);
* Presence of finger pain with a neuropathic pain component (DN4 score ≥ 4/10)
* Inadequate response, adverse reactions, and/or contraindications to conventional analgesics and NSAIDs;

Exclusion Criteria:

* Patient with isolated rhizarthrosis;
* Patient with other joint disease affecting the fingers (gout, chondrocalcinosis, RA, spondyloarthritis, psoriatic arthritis);
* Patient with upper extremity pain syndrome that may interfere with the assessment of finger pain;
* Patient with another pathology responsible for neuropathic hand pain (carpal tunnel syndrome, diabetic neuropathy, Guyon's tunnel syndrome, cervicobrachial neuralgia, brachial plexitis);
* Patient with skin lesions on the fingers (psoriasis, wounds, chronic ulcers, eczema, shingles, dermatitis);
* Patient with poorly controlled high blood pressure;
* Patient with hypersensitivity to capsaicin;
* Patient who had 8% capsaicin patch use in the year prior to the study;
* Patient who has received intramuscular, intra-articular or intravenous corticosteroid therapy, another disease-modifying anti-rheumatic therapy (methotrexate, salazopyrine) or an intra-articular injection into the joints of the fingers within the previous 3 months;
* Patient wearing wrist or finger orthoses in the previous month;
* Patient with fibromyalgia;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-07 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain in the fingers | Day 60
  measured on a visual analogic scale ranging from 0 to 100 mm

SECONDARY OUTCOMES:
Functional disability | Day 60
  Cochin Hand Functional Disability Scale score, Each question is rated from 0 (no difficulty) to 5 (impossible). Total score for 18 questions: 0 - 90. The higher the score, the more impaired the physical function.
Functional index | Day 60
  Modified Functional Index for Hand OsteoArthritis score (FIHOA), Each question is rated from 0 (no difficulty) to 3 (impossible). Total score for the 10 questions: 0 - 30. The higher the score, the greater the functional disability.
Anxiety and depression | Day 60
  Hospital Anxiety and Depression Scale score (HADs), Each question is scored from 0 to 3. Total score for the 7 anxiety or depression questions: 0-21. The higher the score, the more anxious or depressed the patient.
Painful symptoms of osteoarthritis | Day 60
  Osteoarthritis Symptom Inventory Scale score (OASIS9). Localized pain component = 4 questions rated from 0 (no sensation) to 10 (extreme sensation) score = 0-40.
  Neuropathic pain component = 2 questions rated from 0 to 10 score = 0-20. Deep pain component = 3 questions rated from 0 to 10 score = 0-30. Total OASIS score: 0-90. A high score indicates intense pain.
Treatment safety | Day 60
  side effect rate
Patient impression of change | Day 60
  Patient Global Impression of Change " (PGIC) score. The patient evaluates the degree of improvement of his pain
  1. - Strongly improved
  2. - Moderately improved
  3. - Slightly improved
  4. - No change
  5. - Slightly worsened
  6. - Moderately worsened
  7. - Strongly worsened

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Mathieu, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (4):
- France (4):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - HCL Hôpital Edouard Herriot, Lyon
  - AP-HP Hôpital Saint-Antoine, Paris
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan A, Lambert C, Sellam J, Chapurlat R, Marotte H, Pereira B, Thomas T, Tournadre A, Soubrier M, Mathieu S. CADOR (Capsaicin in neuropathic-like pain in digital osteoarthritis) study protocol: a multicentre randomised parallel-group trial. BMJ Open. 2025 Mar 6;15(3):e093409. doi: 10.1136/bmjopen-2024-093409. PMID 40050054